CLINICAL TRIAL: NCT04445129
Title: A Study to Assess the Frequency and Characteristics of Wake and Sleep State Transitions Over Multiple Nights in Subjects With Narcolepsy Type 1 Compared With Healthy Subjects Using a Portable Electroencephalogram Device
Brief Title: Wake and Sleep State Transitions on a Portable Electroencephalogram (EEG) Device in Narcolepsy Type 1 (NT1) and Healthy Participants
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-994-0001; U1111-1251-7993 (Registry Identifier: WHO)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers; Narcolepsy Type 1
MeSH Terms: interventions — Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Narcolepsy Type 1 Participants: Participants with NT1 on stable wake-promoting medications and exclusive of any sleep promoting medications will be fitted with the portable electrocardiogram (ECG) device combined with wrist accelerometry and undergo a 2-night nPSG combined with the portable EEG device.
  Interventions: Device: Portable EEG Device; Device: Portable ECG Device; Device: Accelerometry
- Healthy Participants: Participants who are healthy sex- and age (plus or minus 5 years)-matched controls will be fitted with the portable ECG device combined with wrist accelerometry and undergo a 2-night nPSG combined with the portable EEG device.
  Interventions: Device: Portable EEG Device; Device: Portable ECG Device; Device: Accelerometry

INTERVENTIONS:
Device: Portable EEG Device — Portable EEG device is lightweight and designed for nighttime wear.
Device: Portable ECG Device — Portable ECG device is waterproof and will be adhered to the chest of the participant.
Device: Accelerometry — Portable accelerometry device is noninvasive and will capture data on participant activity level, including intensity of movement, rest, and sleep.

SUMMARY:
The purpose of this study is to determine whether portable devices can provide measurements at home similar to those taken in the clinic, in particular in participant with NT1, and to investigate night-to-night changes in sleep patterns using these devices at home. This study may enable future at-home studies and ultimately lead to a decreased burden on the people who need these measurements.

DETAILED DESCRIPTION:
This is a non-drug study including participants with NT1 and healthy participants using devices designed for at-home assessments. The study will assess whether a portable EEG device provides an EEG signal comparable to inpatient nPSG. The frequency and characteristics of wake and sleep patterns and transitions over multiple nights will also be characterized. Participants with NT1 who will complete the study TAK-994-1501 (NCT04096560) will be eligible to enter the current study following the appropriate washout period (60 days).

The study will enroll approximately 32 participants (16 participants with NT1 and 16 healthy participants). Participants will be enrolled in the 2 groups:

* NT1 Participants
* Healthy Participants

This multi-center trial will be conducted in the United States. The overall time to participate in this study is approximately 8 days. The follow-up visit will occur on Day 10 and during this debrief, participants will answer a questionnaire on user experience (device comfort) for the wearable devices.

ELIGIBILITY:
Inclusion Criteria:

1. Has access to at-home Wi-Fi and can add an internet-ready device with assistance.
2. Body mass index (BMI) between greater than equal to (>=) 18.0 and less than or equal to (<=) 40.0 kilogram per square meter (kg/m^2) at the screening visit.
3. Must have regular sleep-wake habits (example, routinely spending 6.5 to 8.5 hours sleeping nightly, not oversleeping by more than 2 hours on weekends, that is, total sleep not more than approximately 10.5 hours) as determined by investigator interviews and confirmed in accelerometry/actigraphy records obtained between screening and first visit (measured using a minimum of 10 day/night consecutive periods) and who regularly fall asleep between 9:30 PM and 12:00 AM (healthy participants only).
4. Must not require use of sleep aids or must be willing to discontinue use of sleep aids for the duration of the study.
5. Has completed the TAK-994-1501 study, the participant is eligible to enter the current study following the appropriate washout period (60 days).

Participants With NT1 Only:

1. With NT1 who is drug-naïve may also be enrolled.
2. With NT1 must present with subjective sleep complaint.
3. With NT1 must have a diagnosis of NT1, as defined by the International Classification of Sleep Disorders, 3rd edition (ICSD-3) criteria.

Exclusion Criteria:

1. Has a current diagnosis of cancer except for squamous or basal cell skin cancer.
2. Has a nicotine or marijuana dependence that is likely to have an effect on sleep (example, a participant who routinely awakens at night to smoke) and/or an unwillingness to discontinue all smoking and nicotine use during the confinement portions of the study.
3. Cannot maintain stable sleep environment at home, for example, due to young children not yet sleeping through the night or partners with disrupted sleep (example, shift workers).
4. Undergoing current treatment for hepatitis B with interferon.
5. Has a risk of suicide according to endorsement of Item 4 or 5 of the screening visit Columbia Suicide Severity Rating Scale (C-SSRS) or has made a suicide attempt in the previous 6 months.
6. Has medical condition, such as past or current epilepsy, seizure, head injury/trauma, medically significant unstable cardiovascular, pulmonary, hepatic, renal, or gastrointestinal disease, that interferes with a normal sleep pattern or would preclude enrollment in the view of the investigator.
7. Has a lifetime history of major psychiatric disorder, such as bipolar disorder or schizophrenia.
8. As of the screening visit and throughout the study, the participant should not be a chronic caffeine user, as defined by an excessive (greater than [>] 600 milligram [mg]/day) caffeine intake per day.
9. Has a medical disorder (other than narcolepsy), associated with excessive daytime sleepiness. This includes clinically significant obstructive sleep apnea or other sleep disturbances that has a significant impact on daytime sleepiness, confirmed by past PSG data (example, apnea hypopnea index >=10, periodic limb movement disorder index in sleep >=15) or a periodic limb movement disorder arousal index of >=10, or as evaluated on interview at the screening visit. Because nPSG data is obtained on Day 1, participants may be removed from study if they meet the above exclusion at the discretion of the principal investigator. Participants removed under this criterion will be replaced.
10. At the time of screening the participant is being treated with nasal or oro-nasal positive airway pressure for any reason.
11. Is currently being prescribed sodium oxybate or has been off of sodium oxybate for less than 4 weeks.
12. Is using varenicline (Chantix).

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Participants, who maintain a consistent sleep-wake cycle and participants with NT1.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Sleep State Scoring From nPSG and Portable EEG Device | up to 2 Nights
  The concordance between EEG signals obtained from the portable EEG device with nPSG over 2 inpatient night stays will be assessed using data obtained during the inpatient setting from nPSG and a portable EEG device. Scoring of sleep stages occur in 30-seconds epoch based on American Academy of Sleep Medicine (AASM) scoring rules. The output from the nPSG and the portable EEG device will be hand scored for each participant, with the rater assigning 1 of 5 sleep/wake stages to each 30 second epoch 3 stages of non-REM (NREM) sleep (N1, N2, N3), rapid eye movement (REM), and wakefulness (W). The nPSG is a standardized procedure used to assess various sleep parameters, including sleep latency and sleep architecture. nPSG will be used to as the comparator to the portable EEG device.
Stage Shift Index (SSI) as Measured by Standard nPSG and EEG Device on Night 2 | Night 2
  SSI will be measured by standard nPSG and portable EEG device on Night 2 in the clinic. SSI will be calculated as the number of transitions between any wake or sleep stage divided by hours of total sleep time. The summary of the frequency of different stages of sleep transitions can be represented by SSI, which can be used to differentiate healthy participant from those with sleep pathology. The correlation between the SSI as measured by the portable EEG device and by the nPSG will be analyzed for participants with NT1 and healthy controls. The nPSG is a standardized procedure used to assess various sleep parameters, including sleep latency and sleep architecture. nPSG will be used as the comparator to the portable EEG device.

SECONDARY OUTCOMES:
SSI as Measured by Standard nPSG and EEG Device During the Period at Home | Nights 3-7
  SSI will be measured by portable EEG device on nights 3-7 at home. SSI will be calculated as the number of transitions between any wake or sleep stage divided by hours of total sleep time. The summary of the frequency of different stages of sleep transitions can be represented by SSI, which can be used to differentiate healthy participant from those with sleep pathology. The SSI will be analyzed using the intrasubject correlation (intraclass correlation across different nights) in participants with NT1 and healthy participants. The nPSG is a standardized procedure used to assess various sleep parameters, including sleep latency and sleep architecture.
Number of Microsleeps and State Transitions During the Maintenance of Wakefulness Tests (MWTs) | Day 2
  Micro sleeps are defined as appearance of any stage of sleep arising out of wakefulness lasting from 3 seconds to less than or equal to (<=) 15 seconds and assessed on signals obtained from portable EEG device. State transition refers to switch between wake and sleep. MWT is a validated, objective measure used to measure excessive daytime somnolence (EDS) in clinical studies. MWT evaluate a person's ability to remain awake under soporific conditions for a defined period. Wakefulness will be measured indirectly by time to fall asleep using MWT. Four 40-minute trials will be administered (each 4 session 40-minute MWT is considered as complete test). Sleep onset is defined as first epoch of greater than 15 seconds of cumulative sleep in a 30-second epoch. Trials are ended after 40 minutes if no sleep occurs/after unequivocal sleep, defined as 3 consecutive epochs of stage 1 sleep or 1 epoch of any other stage of sleep. If no sleep has been observed, then latency is defined as 40 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Development Center Americas, Inc.
Locations (13):
- United States (13):
  - Stanford School of Medicine, Redwood City, California
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - St Francis Medical Institute, Clearwater, Florida
  - NeuroTrials Research, Inc., Atlanta, Georgia
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Sleep Wake Disorders Center, The Bronx, New York
  - Research Carolina Elite, LLC, Denver, North Carolina
  - CTI Clinical Trial and Consulting Services, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/